CLINICAL TRIAL: NCT01964248
Title: Evaluation of Local Anesthesia Before Arterial Puncture for Blood Gas Analysis Randomized, Control Placebo Study
Brief Title: Local Anesthesia Before Arterial Puncture for Blood Gas Analysis
Acronym: GAEL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RB 12.011 (GAEL)
Record Dates: First submitted 2013-07-25; First posted 2013-10-17 (Estimated); Last update posted 2015-10-16 (Estimated); Status verified 2015-10

CONDITIONS: Indication of Blood Gas Analysis by Radial Artery Blood Sampling
Keywords: Blood gas analysis; Arterial puncture; Local anesthesia; Eutectic mixture; Lidocaïne/prilocaïne cream (5%); Placebo; Pain Intensity Scale; Numerical Rating Scale

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lidocaïne/prilocaïne (Experimental): * Lidocaine/prilocaine eutectic mixture 5% incorporated in a cream base
  * Single dose: 2 grams (one tube of cream)
  * Cream applied 2 hours before blood sample
  Interventions: Drug: lidocaïne/prilocaïne 5%
- Placebo (Placebo Comparator): * Single dose: 2 grams (one tube of cream)
  * Cream applied 2 hours before blood sample
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Placebo cream applied 2 hours before blood sample
  Other Names: Application placebo cream 2 hours before blood sample
  Arms: Placebo
Drug: lidocaïne/prilocaïne 5% — Application cream lidocaïne/prilocaïne (5%) 2 hours before blood sample
  Arms: Lidocaïne/prilocaïne

SUMMARY:
The aim of the study is to evaluate the interest of Local Anesthesia (lidocaïne/prilocaïne versus placebo)before arterial puncture for Blood Gas Analysis. The pain is measured with a numeric Pain Intensity for all patients included.

DETAILED DESCRIPTION:
In an approach of continuous improvement of the quality of the care, this project joins logically after a reflection on the treatment of pain generated by the care in the department of Pneumology 1 / septic Thoracic and vascular Cardiac Surgery.

The arterial puncture for blood gas analysis is an act with aim diagnosis which allows to study gases of the arterial blood to watch the hematosis of the patient. This act appears at the top of the anticipated care as painful by the nursing teams.

In the literature, we find no study carried out with the eutectic mixture lidocaïne prilocaïne. Other local anesthetics and other local ways of administration were estimated and the results diverge as for the efficiency of a local anesthetic for the arterial blood sample at the level radial nerve. Finally authors showed a correlation between certain factors(mailmen) and the painful character of the arterial blood sample, without defining really of population.

In this context, it is necessary to estimate the interest of a local anesthetic before arterial sampling of blood by a study randomized in insu double and versus placebo.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged more than 18 years old, having signed an enlightened consent, who have an indication of gazometry by taking radial nerve
* Patients capable of estimating the pain felt with numeric pain intensity scale
* Patients with numeric pain intensity scale = 0 before sample of blood
* Patients with no contraindication or no allergy of an anesthetic such as lidocaine

Exclusion Criteria:

* Patients aged less than 18 years old
* Patients incapable of estimating the pain felt with numeric pain intensity scale
* Patients with numeric pain intensity scale > 0 before sample of blood
* Patients for whom the arterial taking is impossible for the level radial nerve
* Hypersensibility to local anesthetics of the amide-type or other component of lidocaïne/prilocaïne cream
* Porphyries known
* Pregnant woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2012-12; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
interest of local anesthesia (lidocaïne/prilocaïne) | 1 hour
  Determine the interest of local anesthesia with association of lidocaïne/prilocaïne before arteriel puncture for gas analysis

CONTACTS AND LOCATIONS:
Overall Officials: Francis COUTURAUD, Professor, Principal Investigator — Hôpital Morvan, CHRU de Brest
Locations (1):
- Monocentric study, Brest, France

REFERENCES:
- [Derived] Beaumont M, Goret M, Orione C, Fauche A, Nowak E, Dion A, Darnois V, Tromeur C, Cogulet V, Leroyer C, Couturaud F, Le Mao R. Effect of Local Anesthesia on Pain During Arterial Puncture: The GAEL Randomized Placebo-Controlled Trial. Respir Care. 2021 Jun;66(6):976-982. doi: 10.4187/respcare.08328. Epub 2021 Mar 23. PMID 33758058